CLINICAL TRIAL: NCT04378478
Title: Urological Management of Complications of Penile Constriction Devices: French National Retrospective Study and Literature Review
Brief Title: Urological Management of Complications of Penile Constriction Devices:
Acronym: PCD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0256
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Sexual Dysfunction
Keywords: Penile constriction device; Cockering; Emergency care; Penile strangulation; Urinary dysfunction
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Wearing a penile ring is justified by international societies of Urology (AFU, EAU, AUA) only for the treatment of erectile dysfunction with vacuum. In this case, it is a constriction rubber band that can only be worn for 30 minutes.

Nowadays, wearing a cockring device for recreational purposes can lead to complications secondary to ischemia caused by strangulation of the penis and/or scrotum.

The variety of devices and materials used (metallic and/or alloys in particular) sometimes makes it difficult to remove them, requiring expensive surgery and dedicated equipment.

There is no official recommendation for the management of these complications.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years old
* Peyronie's disease stable for more than 3 months after 12 to 18 months of evolution
* Any patient care for this pathology in public or private healthcare hospitals in France

Exclusion criteria:

- Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient has complications secondary to ischemia caused by strangulation of the penis and / or scrotum
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-11-02 (Actual)

PRIMARY OUTCOMES:
To draw up recommendations for the emergency management of these complications thanks to a study of the (few) cases treated in France and a review of the literature | 1 day
  To draw up recommendations for the emergency management of these complications thanks to a study of the (few) cases treated in France and a review of the literature

SECONDARY OUTCOMES:
Studying | 1 day
  The co-morbidities of these patients (psychiatric pathologies for example)
Studying | 1 day
  The mid- and long-term urinary and sexual functions of these patients

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Fortier, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC